CLINICAL TRIAL: NCT00863954
Title: A Controlled Pilot Study of the Application of Magnetic Fields Using the Resonator in Adjunctive Management of Type 2 Diabetes
Brief Title: Application of Magnetic Fields as Adjunctive Treatment for Type II Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Allen S. Braswell CEO, pico-tesla Magnetic Therapies, LLC, pico-tesla Magnetic Therapies, LLC
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 08165-01
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Output A (Active Comparator)
  Interventions: Device: Resonator Device
- Output B (Active Comparator)
  Interventions: Device: Resonator Device
- Output C (Active Comparator)
  Interventions: Device: Resonator Device
- Output D (Active Comparator)
  Interventions: Device: Resonator Device
- Output E (Active Comparator)
  Interventions: Device: Resonator Device
- Output F (Active Comparator)
  Interventions: Device: Resonator Device

INTERVENTIONS:
Device: Resonator Device — comparison of different parameter settings of electromagnetic fields using the Resonator Device

SUMMARY:
The purpose of this study is to see if using a device called the Resonator, that puts out a very low electromagnetic field, effects blood glucose and A1c levels in people with Type 2 Diabetes.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether application of magnetic fields generated by the Resonator result in statistically significant reductions in finger stick blood glucose levels, serum glucose and hemoglobin A1c levels. The study will also investigate any induced changes in serum lipids and liver function tests as indirect markers of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Type II Diabetes Mellitus with A1c level above the upper limit of normal
* Subject currently performs routine finger stick blood sugar testing
* Subject is ambulatory
* None or stable medication regimen without significant side effects for at least 6 months, willingness and ability to maintain the stable medication regimen throughout the course of the study.
* Hemoglobin A1c levels within a 0.8% range of patient mean A1c level for the last two documented determinations, that must be within 2 years of the baseline testing date.
* Willingness to test finger stick blood sugars according to protocol.
* Willingness to have lab test blood draws performed according to protocol
* Willingness to maintain stable diet and activity regimen for the duration of the study.
* Willing and able to abstain from partaking in any non-essential existing or new treatments to improve serum blood sugar levels.
* Adequate contraceptive measures for female subjects
* Male or female
* Any ethnic group
* Between 21 and 80 years of age

Exclusion Criteria:

* Change in medical regimen within 6 months prior to initiation of study
* Any signs of Type I diabetes
* Active infectious process within 3 weeks of study initiation causing wide fluctuations in finger stick blood sugar level.
* Change in BMI of greater than 6% within a 6 month period prior to study initiation
* Any planned revascularization procedure
* Symptomatic congestive heart failure
* Leg or foot ulceration or open wounds
* Gangrene
* History of intermittent claudication
* Hemodialysis
* Currently being treated for malignancy
* Currently being treated with oral or intravenous catabolic steroids.
* Reported consumption of more than 14 alcoholic drinks per week.
* Pregnant, breast feeding,or planning pregnancy prior to the end of participation.
* Developmental disability or cognitive impairment that would make it difficult for the subject to partake in the clinical study, including adequate comprehension of the informed consent form and ability to record the necessary measurements.
* Uncontrolled hypertension
* Uncontrolled atrial fibrillation or other uncontrolled arrythmias, e.g. tachycardia, bradycardia
* Uncontrolled seizure disorder
* Uncontrolled, unstable, or untreated medical conditions which may significantly impact the subjects health or ability to complete the entire study, in the opinion of the investigator

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Reduction in blood glucose and A1c levels at endpoint compared to start | Start point, 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- pico-tesla Magnetic Therapies, Littleton, Colorado, United States